CLINICAL TRIAL: NCT05724524
Title: Exploratory Study on the Role of the Digestive Microbiota and Bacterial Translocation in the Immune Activation Profile Associated With Insulin Resistance in Male Caucasian Adults Living With HIV-1 on Effective Antiretroviral Therapy.
Brief Title: Exploratory Study on the Role of the Digestive Microbiota in Adults Living With HIV-1
Acronym: MICRACTIVIH
Status: Withdrawn | Type: Observational
Why Stopped: no started
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI GCS-MERRI/2019/JPL-01
Record Dates: First submitted 2022-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum and stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Profile 2: People living with HIV with immune activation profile 2: inflammatory profile - high level of sTNFRI
  Interventions: Other: Stool sample collection; Other: Blood sample collection
- Other profiles: People living with HIV with immune activation profiles1 + 3-5: T8, NK, T4 and monocyte profiles
  Interventions: Other: Stool sample collection; Other: Blood sample collection

INTERVENTIONS:
Other: Stool sample collection — 50mg stool sample taken for protein extraction
Other: Blood sample collection — Venous blood sample taken for analysis of serum and plasma

SUMMARY:
Chronic immune activation present in aviremic people living with HIV under treatment promotes the onset of insulin resistance and metabolic syndrome, paving the way for the comorbidities that are currently the main causes of morbidity. This activation continues despite effective antiretroviral therapy. In the ACTIVIH study (NCT02334943) the analysis of 68 AI markers allowed classification of 120 aviremic PLHIV under treatment for at least 2 years according to 5 different immune activation profiles. Among these 5 profiles, Profile 2 was characterized by high blood pressure figures, high waist sizes, low HDL-cholesterol levels, high triglyceridemia, and especially hyperinsulinemia. Several studies have shown that the digestive microbiota of this population is less rich and less diverse than that of healthy subjects. However, the digestive microbiota and in particular bacterial proteins and metabolites seem to play a key role in immune activation in people living with HIV. Finally, the digestive microbiota has already been shown to have an impact on insulin sensitivity.

The study investigators hypothesize that a particular digestive microbiota could promote the appearance of Profile 2. This microbiota could be the cause of digestive dysbiosis leading to intestinal inflammation, digestive permeability and bacterial translocation.

ELIGIBILITY:
Inclusion Criteria:

* Patient informed of the implementation of the study, its objectives, its constraints and the patient's rights.
* Male and Caucasian patient.
* Patient with HIV-1 infection determined by positive serology or plasma viral load (HIV RNA) measurement.
* Patient on effective triple antiretroviral therapy, stable for more than 6 months, with a plasma viral load <50 copies / ml for at least 6 months before inclusion (2 measurements).
* Patient whose immune activation profile has been characterized beforehand (profiles 1, 2, 3, 4 and 5).
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* Vulnerable person according to article L1121-6 of the CSP.
* Adult person protected according to article L1121-8 of the CSP.
* Patient presenting with a non-infectious pathology which may be the cause of an immune abnormality.
* Patient having undergone treatment with an immunomodulator molecule or chemotherapy within 60 days before inclusion in the research or has an indication planned for the duration of the research.
* Patient with a chronic digestive pathology or who had been operated on the previous year
* The subject is participating in a category 1 interventional study, has participated in another interventional study in the last 3 months or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men with HIV-1 infection on effective antiretroviral therapy stable for more than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Nature of gut microbiota bacterial proteins in patients with immune activation profile 2 versus all other profiles | Day 0
  Number of bacterial proteins present in stool samples from patients, identified by high-performance liquid chromatography mass spectrometry
Nature of gut microbiota taxonomy in patients with immune activation profile 2 versus all other profiles | Day 0
  Number of operational taxonomic units present in stool samples from patients, identified by high-performance liquid chromatography mass spectrometry
Relative quantification of gut microbiota bacterial proteins in patients with immune activation profile 2 versus all other profiles | Day 0
  Percentage of the various bacterial proteins present in stool samples from patients, identified by high-performance liquid chromatography mass spectrometry (%)
Relative quantification of gut microbiota taxonomy in patients with immune activation profile 2 versus all other profiles | Day 0
  Percentage of the various operational taxonomic units present in stool samples from patients, identified by high-performance liquid chromatography mass spectrometry (%)

SECONDARY OUTCOMES:
Richness of Firmicutes and Bacteroidetes in patients with immune activation profile 2 versus all other profiles | Day 0
  Rarefaction curves
Diversity of Firmicutes and Bacteroidetes in patients with immune activation profile 2 versus all other profiles | Day 0
  Shannon index
beta-diversity of Firmicutes and Bacteroidetes in patients with immune activation profile 2 versus all other profiles | Day 0
  Unifrac
Level of phyla and minority species in the stool in patients with immune activation profile 2 versus all other profiles | Day 0
  high-performance liquid chromatography mass spectrometry
Level of CD14S in serum of patients with immune activation profile 2 versus all other profiles | Day 0
  ng/ml by ELISA
Level of Lipopolysaccharide Binding Protein (LBP) in serum of patients with immune activation profile 2 versus all other profiles | Day 0
  pg/ml by ELISA
Level of intestinal fatty acid binding protein (I-FABP) in serum of patients with immune activation profile 2 versus all other profiles | Day 0
  ng/ml by ELISA
Level of bacterial 16S rDNA in plasma of patients with immune activation profile 2 versus all other profiles | Day 0
  Copies/µl
Transcriptomic analysis of peripheral blood mononuclear cells | Day 0
  RNAseq

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Lavigne, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (2):
- France (2):
  - CHU Gui de Chauliac, Montpellier
  - CHU de Nîmes, Nîmes